CLINICAL TRIAL: NCT00192361
Title: A Randomized, Double-Blind Trial of the Safety, Transmissibility, and Phenotypic and Genotypic Stability of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T), in Children Who Attend Day Care. (Final Report Version 2.0)
Brief Title: Trial of the Safety, Transmissibility, and Phenotypic and Genotypic Stability of Influenza Virus Vaccine,(CAIV-T), in Children Who Attend Day Care. (Final Report Version 2.0)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D153 P500
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2006-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
To assess whether CAIV-T was transmitted from vaccinated children to their unvaccinated contacts in a day care setting; and if so, to estimate the rate of transmission.

ELIGIBILITY:
Inclusion Criteria:

* who were at least 8 months and less than 36 months of age (had not reached their 3rd birthday) at the time of enrollment, and in good health as determined by medical history, physical examination, and clinical judgment;
* whose parent or legal guardian had provided written informed consent after the nature of the study had been explained;
* who, along with their parent or legal guardian, were available for the duration of the study (42 days post-vaccination of first study dose or 42 days post-vaccination of supplemental dose of CAIV-T);
* whose parent/legal guardian could be reached by telephone by study staff for the postimmunization contacts;
* who attended day care at least three days per week and four hours per day;
* who was one of at least 4 children in a contact group/playroom (at least 4 children in such a group were required to be randomized in the study).

Exclusion Criteria:

* whose parents or legal guardians were perceived to be unreliable or unavailable for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease and asthma;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there was intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* with an immunosuppressed or compromised individual in the same playroom or living in the same household;
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational);
* with a documented history of hypersensitivity to egg or egg protein;
* with a respiratory illness with wheezing within two weeks prior to enrollment;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for whom use was anticipated during the study;
* who were administered any live virus vaccine within one month prior to enrollment or expected receipt of another live virus vaccine within one month of vaccination in this study;
* who were administered any inactivated vaccine within two weeks prior to enrollment or expected receipt of another inactivated vaccine within three weeks of vaccination in this study;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results.

Ages: 8 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200
Dates: Start 1999-11

PRIMARY OUTCOMES:
The primary endpoint of the study was the determination of the proportion of placebo recipients from whom any of the vaccine strains were isolated.

SECONDARY OUTCOMES:
The endpoint for children who received CAIV-T was the first nasal swab scored positive for viral shedding in
which the vaccine virus phenotype (cold-adapted and temperature sensitive) or genotype (6:2 reassortant) was
not preserved. Genotypic and phenotypic stability were summarized as the proportion of all vaccine viruspositive
isolates which retained the cold-adapted phenotype, temperature-sensitive phenotype or the 6:2
reassortant genotype of the vaccine strains.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- Kauppakatu Clinic, Tampere, Finland